CLINICAL TRIAL: NCT06293755
Title: The Efficacy of Microneedle Patch With Botulinum Toxin in Management of Enlarged Facial Pores Compared to Intradermal Botulinum Toxin
Brief Title: Microneedle Patch With Botulinum Toxin in Management of Enlarged Facial Pores
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dhurakij Pundit University (Other)
Responsible Party: Principal Investigator, Chotip Jitudomtham, Chotip Jitudomtham, Dhurakij Pundit University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: COA022/66
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Enlarged Pores
MeSH Terms: interventions — Injections, Intradermal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedle patch with Botulinum toxin (Experimental): Participants recieve microneedle path with 20 units Botulinum toxin at nose and cheek one side.
  Interventions: Device: Microneedle patch
- Intradermal Botulinum toxin injection (Active Comparator): Participants recieve intradermal 20 units Botulinum toxin injection at nose and cheek in other side.
  Interventions: Device: Intradermal injection

INTERVENTIONS:
Device: Microneedle patch — with 20 units botulinum toxin
  Arms: Microneedle patch with Botulinum toxin
Device: Intradermal injection — with 20 units botulinum toxin
  Arms: Intradermal Botulinum toxin injection

SUMMARY:
The purpose of this study is to assess the efficacy and safety of microneedle patch with botulinum toxin for improving enlarged pores.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and concerned about enlarged pores
* Have pore size 0.3-0.6 mm
* Have pore parameter in each other side of faces not different more than 5%

Exclusion Criteria:

* Any neuromuscular condition
* Pregnancy or breast feeding
* History of allergy : Botulinum toxin, topical anesthesia
* History of keloid or hypertrophic scar
* History of coagulation or receiving medication that causes coagulation disorder
* Using drugs that have interaction with Botulinum toxin
* Using topical medication that improves enlarged pores in 1 month
* Taking medication that improves enlarged pores in 1 month
* Receiving the laser/treatment/chemical peeling in 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-03-05 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of enlarged pores as measured by VISIA (pores parameter) and using pore score | Post-intervention, week 4 and week 16
  the used pore scores, patients with visible pores took the score "1," and those with enlarged pores took "2." When black heads were embedded on facial pores the score was "3." The scores were assessed by 2 investigators who were blinded to the treatment used on each side.

CONTACTS AND LOCATIONS:
Overall Officials: Chotip Jitudomtham, MD, Principal Investigator — Dhurakij Pundit University
Locations (1):
- Dhurakij Pundit University, Lak Si, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salem RM, Salah SAE, Ibrahim SE. Microbotox injection versus its topical application following microneedling in the treatment of wide facial pores: A split face comparative study. J Cosmet Dermatol. 2023 Apr;22(4):1249-1255. doi: 10.1111/jocd.15590. Epub 2023 Jan 6. PMID 36606384